CLINICAL TRIAL: NCT00511836
Title: The Effects of VIVITROL® on Alcohol-Related Cue-Induced Craving and BOLD [Blood Oxygen-level-dependent] Functional Magnetic Resolution Imaging (fMRI) Signal Activation Patterns
Brief Title: ALK21-018: Effects of Medisorb® Naltrexone (VIVITROL®) on Alcohol Craving in Treatment-seeking, Alcohol-dependent Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALK21-018
Record Dates: First submitted 2007-08-02; First posted 2007-08-06 (Estimated); Results first posted 2010-12-07 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Alcohol Dependence
Keywords: alcoholism; addiction; alcohol detoxification
MeSH Terms: conditions — Alcoholism; Behavior, Addictive | interventions — vivitrol; Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- VIVITROL 380 mg (Experimental)
  Interventions: Drug: VIVITROL 380 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VIVITROL 380 mg — Administered via intramuscular (IM) injection once during the double-blind phase and for 2 additional injections, 4 weeks apart, during the optional open-label extension.
  Other Names: naltrexone for extended-release injectable suspension; Medisorb® naltrexone
  Arms: VIVITROL 380 mg
Drug: Placebo — Placebo matching VIVITROL 380 mg was administered by IM injection once during the double-blind phase, only.
  Arms: Placebo

SUMMARY:
This was a study of the effects of VIVITROL® on alcohol cue-induced craving and the associated brain activation patterns in alcohol-dependent adults who had recently completed alcohol detoxification and were seeking further treatment for their alcohol dependence. The study was powered to to detect whether VIVITROL attenuates or blocks the BOLD signal increases in response to alcohol-related cues.

In the double-blind portion, subjects received a single administration of study drug (VIVITROL 380 mg or placebo). Subjects who completed the double-blind portion could opt to continue to the open-label portion and receive 2 additional months of treatment with VIVITROL 380 mg.

DETAILED DESCRIPTION:
The double-blind phase consisted of 6 visits over a 5- to 6-week period and included 2 telephone contacts and 2 functional magnetic resonance imaging (fMRI) scans.

The optional open-label extension included 2 visits approximately 1 month apart. Subjects who completed both phases participated in a total of 8 scheduled visits (including 2 fMRI scans and 2 telephone contacts) over a period of up to 14 weeks.

At screening, eligible, consenting subjects were given an Actiwatch®-Score device. They were instructed to record their alcohol craving using this device throughout the double-blind phase. The Actiwatch was programmed to beep every 3 hours ±20 minutes, thereby signaling the subjects to enter their craving or desire to use alcohol, at that exact moment, on a scale of 0 to 10 (with 0 being no craving at all and 10 being extreme craving). In addition, subjects entered any drug and/or alcohol use at the time of occurrence. The Actiwatch was not utilized in the open-label portion of the study.

ELIGIBILITY:
Primary Inclusion Criteria:

* Current diagnosis of alcohol dependence, meeting at least 3 criteria from the Diagnostic and Statistical Manual of Mental Disorders, 4th Ed. (DSM-IV)
* Recently completed alcohol detoxification and seeking treatment for alcohol dependence
* Women of childbearing potential must agree to use an approved method of contraception for study duration

Primary Exclusion Criteria:

* Pregnancy or lactation
* Evidence of hepatic failure including: ascites, bilirubin >10% above upper limit of normal (ULN) and/or esophageal variceal disease
* Current dependence (within the past year) to benzodiazepines or cocaine, or current or history of opioid dependence according to DSM-IV criteria
* Use of any opioids and/or methadone within 14 days prior to the screening visit, or likely to require opioid therapy during the study period
* Previous enrollment in a VIVITROL clinical trial or previous VIVITROL experience
* Known intolerance and/or hypersensitivity to naltrexone, carboxymethylcellulose, or polylactide-co-glycolide (PLG)
* Parole, probation, or pending legal proceedings having the potential for incarceration during the study period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-07; Primary Completion 2009-06 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott E. Lukas, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

REFERENCES:
- [Result] Lukas SE, Lowen SB, Lindsey KP, Conn N, Tartarini W, Rodolico J, Mallya G, Palmer C, Penetar DM. Extended-release naltrexone (XR-NTX) attenuates brain responses to alcohol cues in alcohol-dependent volunteers: a bold FMRI study. Neuroimage. 2013 Sep;78:176-85. doi: 10.1016/j.neuroimage.2013.03.055. Epub 2013 Apr 6. PMID 23571420

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at a single clinical study center. The first subject was enrolled in July 2007. The last subject was enrolled in May 2009.
Pre-assignment Details: Screening evaluations were conducted during a 1-week period. All screening evaluations were to be completed at least 2 days before randomization and dosing.
Groups:
- VIVITROL 380 mg: VIVITROL 380 mg (naltrexone for extended-release injectable suspension) - single administration via intramuscular (IM) injection on Day 1
- Placebo: Placebo matching VIVITROL 380 mg - single administration via intramuscular injection on Day 1
Period: Double-blind Period
Arm/Group | VIVITROL 380 mg | Placebo
Started | 16 | 15
Completed | 15 | 15
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Optional Open-label VIVITROL (2 Months)
Arm/Group | VIVITROL 380 mg | Placebo
Started | 22 (Subjects who received placebo during Month 1 switched to VIVITROL for the optional extension phase.) | 0 (Not all subjects from the double-blind phase entered the optional open-label extension.)
Completed | 6 | 0
Not Completed | 16 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VIVITROL 380 mg | Placebo | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 15 | 31
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.3 (8.8) | 44.8 (9.5) | 46.6 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 11 | 10 | 21
Region of Enrollment [Number; unit: participants]
  United States | 16 | 15 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Blood Oxygen-level-dependent (BOLD) Signal Activation Values Detected in the Reward Circuitry of the Brain in Alcohol-dependent Subjects After Presentation of Alcohol-related Cues.
Description: As was standard among fMRI studies conducted at the study site at the time, a change in BOLD signal in the range of 5% to 6% in anterior cingulate as measured using a 3T magnet,is considered highly significant in block-designed experiments.
Time Frame: 14 days (Baseline to Day 14)
Population: Analyses include all randomized, dosed subjects who had functional magnetic resolution imaging (fMRI) on Day 14. No data were imputed.
Measure: Mean (Standard Deviation); unit: Percentage (%) of Change
Arm/Group | VIVITROL 380 mg | Placebo
Number analyzed (Participants) | 15 | 13
Percentage (%) of Change | 0.041 (0.036) | -0.044 (0.049)
Statistical Analysis 1: Comparison: VIVITROL 380 mg vs Placebo; Null hypothesis: mean treatment difference=0; Test type: Superiority or Other; p < 0.00002, t-test, 1 sided

2. Secondary Outcome: Change From Baseline in Obsessive-Compulsive Drinking Scale (OCDS) Score in Alcohol-dependent Subjects
Description: There are 14 items on the Obsessive Compulsive Drinking Scale (OCDS). The scale is scored from 0 to 40 (units). A score of 0 units indicates no obsession-compulsion with respect to alcohol (best score). A score of 40 units indicates maximum obsession-compulsion with respect to alcohol (worst score). A negative Change from Baseline value indicates an improvement. For scoring methods, see: Anton RF, Moak DH, Latham P (1995), The Obsessive Compulsive Drinking Scale: A self-rated instrument for the quantification of thoughts about alcohol and drinking behavior. Alcohol Clin Exp Res 19:92-9.
Time Frame: 28 days (Baseline to Day 28)
Population: All randomized subjects who received at least 1 dose of study drug and had an Obsessive-Compulsive Drinking Scale (OCDS) assessment at Day 28 were included in this analysis. No last-observation-carried-forward (LOCF) approach was used.
Measure: Mean (Standard Deviation); unit: Change in OCDS score
Arm/Group | VIVITROL 380 mg | Placebo
Number analyzed (Participants) | 15 | 15
Change in OCDS score | -8.5 (5.7) | -7.3 (6.4)

3. Secondary Outcome: Change From Baseline in Daily Craving Score in Alcohol-dependent Subjects (Actiwatch Data)
Description: The Actiwatch-Score device (MiniMitter Co.) was used to collect data on daily alcohol craving. The Actiwatch device is a wrist-worn, battery-operated monitor programmed to beep every 3 hours ±20 minutes, to signal the subjects to enter their alcohol craving or desire to use alcohol at that exact moment on a scale of 0 to 10 units: 0 indicates no craving at all (best score) and 10 indicates extreme craving (worst score). A negative result for Change in Baseline at Day 28 indicates an improvement in daily craving as of 1 month after study drug administration.
Time Frame: 28 days (Baseline to Day 28)
Population: All randomized subjects who received at least 1 dose of study drug and had a craving score assessment at Day 28 were included in this analysis. No last-observation-carried-forward (LOCF) approach was used.
Measure: Mean (Standard Deviation); unit: Change in Daily Craving Score
Arm/Group | VIVITROL 380 mg | Placebo
Number analyzed (Participants) | 14 | 15
Change in Daily Craving Score | -0.846 (0.881) | -0.789 (0.986)

4. Primary Outcome: Change From Baseline in BOLD Signal Activation Values for the Inferior Frontal Gyrus
Time Frame: 14 days (Baseline to Day 14)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage (%) of Change
Arm/Group | VIVITROL 380 mg | Placebo
Number analyzed (Participants) | 15 | 13
Percentage (%) of Change | 0.001 (0.055) | -0.067 (0.078)
Statistical Analysis 1: Comparison: VIVITROL 380 mg vs Placebo; Null hypothesis: mean treatment difference=0; Test type: Superiority or Other; p < 0.013, t-test, 1 sided

5. Primary Outcome: Change From Baseline in BOLD Signal Activation Values in the Reward Circuitry
Time Frame: 14 days (Baseline to Day 14)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage (%) of Change
Arm/Group | VIVITROL 380 mg | Placebo
Number analyzed (Participants) | 15 | 13
Percentage (%) of Change | -0.018 (0.105) | -0.060 (0.074)
Statistical Analysis 1: Comparison: VIVITROL 380 mg vs Placebo; Null hypothesis: mean treatment difference=0; Test type: Superiority or Other; p = 0.245, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: From the time of consent, adverse events (AEs) were monitored continuously in each subject until 30 days after his or her last administration of study drug.
Description: In the open-label period, VIVITROL was administered in an unblinded manner to subjects who chose to continue in this optional extension; there was no control group in the open-label phase.
Groups:
- VIVITROL 380 mg (Double-blind Period): VIVITROL 380 mg (naltrexone for extended-release injectable suspension). Data are described for the initial 28-day double-blind period.
- Placebo (Double-blind Period): Placebo for VIVITROL 380 mg. Data are described for the initial 28-day double-blind period.
- Optional Open-label VIVITROL Period (2 Months): Following the 28-day, double-blind treatment period, all subjects were offered a chance to receive open-label VIVITROL for an additional 2 months (2 injections, each separated by 1 month). Safety data are described for all subjects in the VIVITROL open-label period, regardless of the treatment received (VIVITROL or placebo) for the first month.
Arm/Group | VIVITROL 380 mg (Double-blind Period) | Placebo (Double-blind Period) | Optional Open-label VIVITROL Period (2 Months)
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15 | 0/22
Other Adverse Events (participants affected / at risk) | 6/16 | 10/15 | 7/22
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VIVITROL 380 mg (Double-blind Period) (N=16) | Placebo (Double-blind Period) (N=15) | Optional Open-label VIVITROL Period (2 Months) (N=22)
Injection site pain (General disorders) | 1 | 3 | 0
Injection site induration (General disorders) | 2 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Injection site abcess (General disorders) | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 3 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 1
Abnormal dreams (Psychiatric disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Euphoric mood (Psychiatric disorders) | 1 | 0 | 0
Irritability (General disorders) | 0 | 1 | 0
Libido decreased (Psychiatric disorders) | 0 | 1 | 0
Sexual dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 0 | 1
Hallucinations, visual (Psychiatric disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 3 | 1
Fatigue (General disorders) | 0 | 1 | 1
Pain (General disorders) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Ear congestion (Ear and labyrinth disorders) | 1 | 0 | 0
Chest x-ray abnormal (Investigations) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Blood alkaline phosphate increased (Investigations) | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1
Haematemesis (Vascular disorders) | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The study was powered to detect whether VIVITROL blocks the fMRI BOLD signal increase in response to alcohol-related cues as compared to placebo. Results of the secondary endpoints should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI/Institution may publish study results for noncommercial purposes. Sponsor will have 30 days to review a proposed publication. PI/Institution will delete any Sponsor Confidential Information other than study results, will revise a publication based on regulatory requirements of Sponsor as manufacture of the study drug, and will delay publication for no more than 60 days to allow for filing of patent applications to protect Sponsor's intellectual property contained in such publication.